CLINICAL TRIAL: NCT04104152
Title: CSD190203: A Study to Determine Subject Puffing Patterns of an Electronic Nicotine Delivery System in an Ambulatory Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CSD190203
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Smoking; Smoking Behaviors; Tobacco Use; Tobacco Smoking
MeSH Terms: conditions — Smoking; Tobacco Use; Tobacco Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ENDS 2.4% nicotine (Experimental): Subjects will be assigned to one of four flavors variants of 2.4% ENDS products based on their preferred UB flavor.
  Interventions: Other: CSD1902-11; Other: CSD1902-12; Other: CSD1902-13; Other: CSD1902-14
- ENDS 5.0% nicotine (Experimental): Subjects will be assigned to one of four flavors variants of 5.0% ENDS products based on their preferred UB flavor.
  Interventions: Other: CSD1902-21; Other: CSD1902-22; Other: CSD1902-23; Other: CSD1902-24

INTERVENTIONS:
Other: CSD1902-11 — A 2.4% nicotine ENDS product
  Arms: ENDS 2.4% nicotine
Other: CSD1902-12 — A 2.4% nicotine ENDS product
  Arms: ENDS 2.4% nicotine
Other: CSD1902-13 — A 2.4% nicotine ENDS product
  Arms: ENDS 2.4% nicotine
Other: CSD1902-14 — A 2.4% nicotine ENDS product
  Arms: ENDS 2.4% nicotine
Other: CSD1902-21 — A 5.0% nicotine ENDS product
  Arms: ENDS 5.0% nicotine
Other: CSD1902-22 — A 5.0% nicotine ENDS product
  Arms: ENDS 5.0% nicotine
Other: CSD1902-23 — A 5.0% nicotine ENDS product
  Arms: ENDS 5.0% nicotine
Other: CSD1902-24 — A 5.0% nicotine ENDS product
  Arms: ENDS 5.0% nicotine

SUMMARY:
This study will be a single-center, randomized, controlled, open-label, parallel 2-cohort study to evaluate the puffing patterns of individuals switching from a similar usual brand (UB) Electronic Nicotine Delivery System (ENDS) product to either a 2.4% or 5% nicotine level ENDS product in healthy adult ENDS users. This study will be conducted for potential submission to the US Food and Drug Administration (FDA) Center for Tobacco Products (CTP) as part of a Premarket Tobacco Product Application (PMTA) for an Electronic Nicotine Delivery System (ENDS), comprised of an electrical power unit and four flavor variants each with two different levels of nicotine (2.4% and 5.0%).

DETAILED DESCRIPTION:
Potential subjects will complete a pre-screening interview and a Screening Visit to assess their eligibility and, based on meeting eligibility requirements, will be enrolled into the study on the same day of the Screening Visit.

Once enrolled, the subjects will be randomized to either the 5.0% nicotine ENDS products or the 2.4% nicotine ENDS products. Once randomized to the nicotine level, subjects will be assigned to one of the four flavor variants based on alignment with their preferred UB flavor.

Subjects will be provided an orientation to the product and the Product Use and Behavior (PUB) instrument and provided with enough cartridges (sufficient for three weeks of product use [125% their reported weekly use of their UB]) to last the 3-week period of the study.

The subjects will take the products home and use them ad libitum for a 1-week acclimation period followed by a 2-week product use period. During this time product use will be captured by the PUB instrument and their data uploaded to the cloud regularly.

At the conclusion of the 3-week ambulatory period, the subject will return to the clinic, return the ENDS power unit, used and unused ENDS cartridges, and the PUB instrument (and all cables/charger), have his/her health status reevaluated, complete the Product Evaluation Scale (PES) questionnaire and will then be discharged from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and willing to sign an informed consent form (ICF) and complete questionnaires written in English.
2. Generally healthy male or female, 21 to 60 years of age, inclusive, at the time of consent.
3. Positive urine cotinine test at Screening.
4. Non-cylindrical, cartridge-based, closed system, ENDS are the primary form (> 50% of total use over the last month) of tobacco- or nicotine-containing product used within 30 days of Screening.
5. Must have purchased and used 2 or more cartridges per week over the last 30 days. Brief periods of abstinence due to illness, quit attempt (prior to 30 days of Screening), or clinical study participation (prior to 30 days of Screening) will be allowed at the discretion of the Principal Investigator (PI).
6. Primary flavor preference (75% use per week, self-reported) must be either Tobacco, Mint/Menthol, or a Fruit/Berry flavor and listed in the acceptable UB product guide.
7. Females must be willing to use a form of contraception acceptable to the PI from the time of signing the ICF until the end of the study.
8. Must be willing to use a the assigned non-cylindrical, cartridge-based product and only the assigned flavor as their exclusive source of ENDS use for the full duration of the 3-week ambulatory period.
9. Must have a modern IOS/Android phone (as described in the study procedures manual) that allows for both Bluetooth connectivity and internet connectivity and be willing to keep both active for the length of the study.
10. Must be willing to install an application onto their personal smartphone and keep the application active for the length of the study.

Exclusion Criteria:

1. Presence of clinically significant uncontrolled cardiovascular, pulmonary, renal, hepatic, endocrine, gastrointestinal, psychiatric, hematological, neurological disease, or any other concurrent disease or medical condition that, in the opinion of the PI, makes the study participant unsuitable to participate in this clinical study.
2. History or presence of diabetes.
3. Systolic blood pressure of > 160 mmHg or a diastolic blood pressure of > 95 mmHg, measured after being seated for five minutes, with exceptions at the PI's discretion.
4. Scheduled treatment for asthma currently or within the past consecutive 12 months prior to the Screening-Enrollment Visit. As-needed treatment, such as inhalers, may be included at the PI's discretion pending approval from the Medical Monitor.
5. Any history of cancer, except for primary cancers of skin such as localized basal cell/squamous cell carcinoma that has been surgically and/or cryogenically removed.
6. Use of any medication or substance that aids in smoking cessation, including but not limited to any nicotine replacement therapy (NRT, e.g., nicotine gum, lozenge, patch), varenicline (Chantix®), bupropion (Wellbutrin®, Zyban®), or lobelia extract within (≤) 30 days prior to the signing of informed consent.
7. Participation in another clinical trial within (≤) 30 days prior to signing the ICF. The 30-day window for each subject will be derived from the date of the last study event in the previous study to the time of signing the ICF in the current study.
8. Females who have a positive pregnancy test, are pregnant, breastfeeding, or intend to become pregnant during the course of the study.
9. Individuals ≥ 35 years of age currently using systemic, estrogen-containing contraception or hormone replacement therapy.
10. A positive urine drug screen without evidence of prescribed corresponding concomitant medication(s) at Screening.
11. Postpones a decision to quit using tobacco- or nicotine-containing products in order to participate in this study or a previous attempt within (≤) 30 days prior to the signing of the ICF.
12. Drinks more than 21 servings of alcoholic beverages per week or has a positive alcohol breathalyzer result at Screening.
13. Determined by the PI to be inappropriate for this study.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 146 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Arithmetic Mean | 2 weeks
  Arithmetic Mean puff duration for 5.0% nicotine and 2.4% nicotine ENDS products across the final two weeks of data collection

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Smith, PhD, Study Director — RAIS
Locations (1):
- High Point Clinical Trials Center, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No